CLINICAL TRIAL: NCT04814134
Title: The STOP-ADHF Study: Stimulation of the Cardiopulmonary Nervous System in Acute Decompensated Heart Failure
Brief Title: Cardionomic STOP-ADHF Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardionomic Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLN-1051-001
Record Dates: First submitted 2021-03-10; First posted 2021-03-24 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Neurostimulation; Contractility; Right Pulmonary Artery
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled in CPNS treatment arm or to the control arm. Treatment with CPNS system includes endovascular stimulation of the cardiac autonomic nerves in addition to standard of care. Subjects in the control arm will receive the available standard treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- CPNS Therapy (Experimental): Treatment with CPNS system: Endovascular stimulation of the cardiac autonomic nerves in addition to standard of care
  Interventions: Device: CPNS Therapy; Other: Standard of care
- Standard of Care (Other): Available standard treatment
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: CPNS Therapy — Endovascular stimulation of the cardiac autonomic nerves in addition to standard of care
  Arms: CPNS Therapy
Other: Standard of care — Available standard treatment

SUMMARY:
STOP-ADHF Study: An evaluation of the safety and performance of the Cardionomic Cardiac Pulmonary Nerve Stimulation (CPNS) system in patients with acute decompensated heart failure.

DETAILED DESCRIPTION:
The STOP-ADHF is a prospective, two-arm, multi-center study to evaluate the safety and performance of the CPNS System in patients with acute decompensated heart failure (ADHF).

The CPNS System is a neuromodulation system, intended to provide acute (≤5 days) endovascular stimulation of the cardiac autonomic nerves in the right pulmonary artery. The system consists of a temporary neuromodulation stimulator catheter and a stimulator.

Approximately 90 patients will be enrolled in the study and will be followed up through 6-months post-discharge from the hospital. Patients enrolled in the treatment group will receive CPNS therapy and followed closely in an intensive care unit setting. Patients enrolled in the control arm in will receive standard treatment for their heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to hospital with a principal diagnosis of ADHF
* BMI adjusted BNP ≥ 500 pg/mL or NT-proBNP ≥ 2000 pg/mL
* LVEF ≤ 50%
* At least one sign or symptom of fluid overload despite the administration of IV furosemide (or equivalent) (at least 40 mg or equivalent)

Exclusion Criteria:

* Received a high dose inotrope or Levosimendan during current hospitalization or treatment with a low dose inotriope within 24 hours before enrollment
* Requires mechanical support
* Cardiogenic shock or impending cardiogenic shock
* Systolic blood pressure < 80mmHg or > 140mmHg
* Symptomatic hypotension
* eGFR < 25 mL/min/1.732

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-09-24 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
Safety Measures | 6 months
  The occurrence of all system and/or procedure related adverse events and serious adverse events and deaths

CONTACTS AND LOCATIONS:
Locations (15):
- United States (9):
  - St. Vincent Hospital, Indianapolis, Indiana
  - Summa Health, Akron, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - University Hospitals, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oklahoma Heart Hospital South, Oklahoma City, Oklahoma
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - Medical City Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
- Belgium (3):
  - OLV Ziekenhuis, Aalst
  - AZ Sint-Jan Brugge, Bruges
  - Antwerp University Hospital, Edegem
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - St. Antonius Ziekenhuis, Nieuwegein
- Punta Pacifica, Panama City, Panama